CLINICAL TRIAL: NCT05128318
Title: Study of the Tumor-adipose Tissue Dialogue: Role of Tumor Acidosis in the Induction of Adipocyte Lipolysis
Brief Title: TuLip : Role of the Tumor Environment in Cancer-related Fat Loss
Acronym: TuLip
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited number of recruited patients
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TuLip
Record Dates: First submitted 2021-10-14; First posted 2021-11-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Cachexia; Adipose Tissue
MeSH Terms: conditions — Neoplasms; Cachexia | interventions — Fundoplication; Cholecystectomy

STUDY DESIGN:
Intervention Model Description: Collection of subcutaneous and visceral adipose tissue from patients with BMI < 30 kg/m2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with BMI < 30 kg/m2 (Experimental): Collection of subcutaneous and visceral adipose tissue pieces of 1-2 cm3 during abdominal surgery procedures
  Interventions: Procedure: Nissen Fundoplication, cholecystectomy

INTERVENTIONS:
Procedure: Nissen Fundoplication, cholecystectomy — Collection of adipose tissue pieces in the context of programmed abdominal surgery to treat to treat hiatal hernia, gastroesophageal reflux or vesicular lithiasis. During the surgery treatment, adipose tissue of 1-2 cm3 will be collected for the protocol by laparoscopy by the surgeon in charge of the procedures.

SUMMARY:
Cancer cachexia is defined as a weight loss of more than 5% over the last 6 months, a loss of body fat and muscle atrophy. It is found in 80% of patients with advanced cancer. In this context, white adipose tissue is a particularly interesting target since its depletion precedes the loss of muscle mass, and is sufficient to induce a decrease in the response to anti-cancer treatments and in the survival of patients.

This cachexia is associated with advanced tumors that present acidosis and metastasis. In this clinical study the investigators would like explore the acid environment effect on the human adipose tissue depletion and more specifically on adipocyte lipolysis.

The main objective of the "TuLip" clinical study is therefore to validate in human subcutaneous and visceral adipocytes that factors secreted by tumor cells cultivated in acid tumor environment stimulate the release of lipids from adipose tissue. Adipocytes retrieves from this study will also be used to validate identified potential lipolytic factors derived from these cells.

DETAILED DESCRIPTION:
This study is a monocentric clinical study. Patients with BMI < 30 kg/m2 will be recruited in the context of programmed abdominal surgery. In this context, subcutaneous and visceral adipose tissue pieces (1-2 cm3) will be collected to explore the lypolytic response of adipocytes ex-vivo to factors secreted by human cancer cell lines.

ELIGIBILITY:
Inclusion Criteria:

* Programmed surgeries in the abdominal area in the Department of Surgery and Transplantation at Cliniques Universitaires Saint-Luc under the supervision of Prof. Dr. Benoit Navez.
* Hospitalization in the context of surgery
* Caucasian
* Age between 18 and 60 years (included).
* Body mass index less than 30 and greater than or equal to 18.5
* Programmed Nissen fundoplication (to treat hiatal hernia and gastroesophageal reflux) or cholecystectomy (to treat vesicular lithiasis), eventration, or parietal surgery .
* Adults capable of expressing their wishes.
* Understanding French

Exclusion Criteria:

* Body mass index below 18.5 and above 30.
* Patients with cancer, infection, autoimmune or inflammatory disease, metabolic syndrome.
* Patients with beta-blockers, hypoglycemics, anti-diabetics, hypolipidemics.
* Adults unable to express their will.
* Not understanding French
* Patients participating in a clinical trial for a drug treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of the lipolytic response of adipocytes isolated from human visceral and subcutaneous adipose tissue to factors derived from cancer cells in acid environment by the glycerol measurement | Up to 100 days after the adipose tissue collection"
  Measure ex-vivo of the lipolysis of subcutaneous and visceral adipocytes in the presence of factors derived from cancer cells. The lipolysis will be assessed by the measure of glycerol (in mol/L) released by adipocytes.
Evaluation of the lipolytic response of adipocytes isolated from human visceral and subcutaneous adipose tissue to factors derived from cancer cells in acid environment by the fatty acid measurement. | Up to 100 days after the adipose tissue collection"
  Measure ex-vivo of the lipolysis of subcutaneous and visceral adipocytes in the presence of factors derived from cancer cells. The lipolysis will be assessed by the measure of free fatty acids (in mol/L) released by adipocytes.

SECONDARY OUTCOMES:
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by western-blot | Up to 2 years after the adipose tissue collection
  Protein analyses by western-blot (arbitrary units).
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by ELISA | Up to 2 years after the adipose tissue collection
  Protein analyses by ELISA (mol/L or g/L).
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by proteomic analyses | Up to 2 years after the adipose tissue collection
  Protein analyses via proteomic analyses (relative units).
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by biochemical analyses | Up to 2 years after the adipose tissue collection
  Biochemical analyses (biochemical kits)
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by metabolomic analyses | Up to 2 years after the adipose tissue collection
  Metabolomic analyses (arbitrary units or mol/L)
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by RNA sequencing | Up to 2 years after the adipose tissue collection
  Measurement of gene expression by RNA sequencing (in counts) of RNA extracted from these ex-vivo cultured human adipocytes.
Evaluation of the lipid metabolism, of adipocytes isolated from human visceral and subcutaneous adipose tissues to factors derived from cancer cells in acid environment, by RT-qPCR | Up to 2 years after the adipose tissue collection
  Measurement of gene expression by RT-qPCR (in relative units) of RNA extracted from these ex-vivo cultured human adipocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Navez, Professor, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lefevre C, Thibaut MM, Loumaye A, Thissen JP, Neyrinck AM, Navez B, Delzenne NM, Feron O, Bindels LB. Tumoral acidosis promotes adipose tissue depletion by fostering adipocyte lipolysis. Mol Metab. 2024 May;83:101930. doi: 10.1016/j.molmet.2024.101930. Epub 2024 Apr 1. PMID 38570069